CLINICAL TRIAL: NCT03326388
Title: A Paediatric Phase I/II Study Of Intermittent Dosing Of The Mek-1 Inhibitor Selumetinib In Children With Neurofibromatosis Type-1 And Inoperable Plexiform Neurofibroma And/Or Progressive Optic Pathway Glioma
Brief Title: Intermittent Dosing Of Selumetinib In Childhood NF1 Associated Tumours
Acronym: INSPECT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15Hi53
Record Dates: First submitted 2017-09-08; First posted 2017-10-31 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Neurofibromatosis Type 1; Plexiform Neurofibroma; Optic Nerve Glioma
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform; Optic Nerve Glioma | interventions — AZD 6244

STUDY DESIGN:
Intervention Model Description: Single Arm Study of Intermittent Schedule of Drug Dosing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selumetinib Intermittent Dosing (Experimental): Phase 1 of the study to evaluate Intermittent Dosing (Selumetinib given twice daily on 5 out of 7 days) in children with NF1 and inoperable plexiform neurofibromas. The Maximum tolerated dose will define the Recommended phase 2 dose of selumetinib.
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — Selumetinib Intermittent Dosing
  Other Names: AZD6244,; ARRY-142886; AR00142886; AR-142886-X

SUMMARY:
Phase I and II study of the MEK inhibitor Selumetinib given twice daily on 5 out of 7 days in children with NF1 and inoperable plexiform neurofibromas or progressive/relapsed optic pathway gliomas.

This study will test the early and late toxicities of selumetinib when it is given in this intermittent schedule (in 5 out of 7 days) and will also test the effectiveness of the drug in reducing the size of plexiform neurofibromas and optic pathway gliomas in children with NF1. It will also test the effectiveness of the drug in improving the participants function in day to day life.

DETAILED DESCRIPTION:
Neurofibromatosis type 1 (NF1) is a common autosomal dominant, progressive disorder with an incidence of 1 in 3,500 of the population. NF1 is characterized by diverse, progressive cutaneous, neurological, skeletal and neoplastic manifestations with no standard drug treatment options available. Patients with NF1 have an increased risk of developing tumours of the central and peripheral nervous system including plexiform neurofibromas (PN) (27%) and optic gliomas (15-20%).

Genetic aberrations targeting the Ras-mitogen-activated protein kinase (MAPK) signalling pathway are a hallmark molecular feature of Low Grade Gliomas (including optic pathway gliomas) and NF1 as well as some low-grade glial-neuronal tumours. The gene responsible for NF1 has been cloned and encodes a protein called neurofibromin. Loss of Neurofibromin is associated with elevated levels of Ras, and Activated Ras results in the initiation of a cascade of signalling events such as activation of Raf and MAPK that leads to increased cell proliferation. Thus MAPK inhibitors offer an attractive novel therapeutic option for both NF1 related PN and optic pathway gliomas

This study will comprise 2 phases. Phase 1 will be a dose escalation phase, designed to establish the correct dose of selumetinib. Phase 1 will be open to NF-1 participants, aged 3 to ≤18 years with inoperable plexiform neurofibromas (PN). This phase of the study will investigate a new intermittent schedule of oral administration of selumetinib, (given twice daily on 5 out of every 7 days) to determine the maximum tolerated dose (MTD) and a recommended phase 2 dose. The starting dose level will be 25mg/m2/dose given twice daily. This was the MTD determined by the Paediatric Brain Tumour Consortium study of Selumetinib in children with NF1 related LGG and the National Cancer Institute study of children with NF1 inoperable PN. In both of these trials selumetinib was given twice daily, every day. The purpose of this phase 1 study will allow the investigators to define the acute and chronic toxicities and pharmacokinetics (PK) of Selumetinib in this population and contribute to determining the effect of Selumetinib on the growth rate of PN.

The Phase 2 part of the study will be a dose expansion study and will be open to 2 groups of participants. Those with progressive NF-1 related optic pathway gliomas (OPG), and those with NF1 related inoperable PN. This part of the study will only commence when the recommended phase 2 dose is established from part 1. The purpose of this part of the study is to determine the effectiveness of the 5 out of 7 day intermittent dosing schedule of Selumetinib, using response rates (and duration of response), appropriate MRI criteria and functional assessments (REINs criteria). The investigators plan to further evaluate the acute and chronic toxicities of selumetinib in this population and to assess the clinical status and quality of life in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age Phase I: ≥3 years and ≤18 years of age at the time of study enrolment, if able to swallow whole capsules.

   Age Phase II: ≥3 years and ≤ 18 years. BSA ≥ 0.55 m2, if able to swallow whole capsules.
2. Diagnosis: Phase I (Dose escalation): Patients with NF1 and inoperable PNs defined as PNs that cannot be surgically completely removed without risk for substantial morbidity due to: encasement of or close proximity to vital structures, invasiveness, or high vascularity of the PN. The PN has to cause morbidity or have the potential to cause significant morbidity, such as (but not limited to) head and neck lesions that could compromise the airway or great vessels, brachial or lumbar plexus lesions that could cause nerve compression and loss of function, lesions that could result in major deformity (e.g., orbital lesions) or are significantly disfiguring, lesions of the extremity that cause limb hypertrophy or loss of function, and painful lesions.

   Histological confirmation of tumour is not necessary in the presence of consistent clinical and radiographic findings, but should be considered if malignant degeneration of a PN is clinically suspected.

   Phase 2 (Dose expansion): Two cohorts are eligible for inclusion in the dose expansion cohort.

   Cohort A (10 subjects) Subjects with NF1 and inoperable PNs (as per Phase I) and Cohort B (10 subjects) Subjects with NF-1 related progressive optic pathway glioma are eligible if the subject has evidence of either clinical (e.g. worsening visual function as per REiNS) or MRI based significant radiological progression and has had at least two lines of standard therapy.

   In addition, all study subjects (phase I and II) must have either positive genetic testing for NF1 from a certified laboratory or have at least one other diagnostic criterion for NF1 listed below:
   * Six or more café-au-lait macules (≥0.5cm in prepubertal subjects or ≥1.5 cm in post pubertal subjects)
   * Freckling in axilla or groin
   * Optic glioma
   * Two or more Lisch nodules
   * A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
   * A first-degree relative with NF1
3. Measurable disease (PN): Subjects must have at least one measurable PN, defined as a lesion of at least 3 cm measured in one dimension. Subjects who underwent surgery for resection of a PN are eligible provided the PN was incompletely resected and is measurable. Measurable disease (OPG): Subjects must have one measurable OPG lesions according to RANO 1.1 i.e. Tumour ≥10 x10mm in maximal perpendicular dimensions on an axial image on MRI with ≤5 mm reconstruction interval.
4. Prior Therapy: Subjects with NF1 will only be eligible if complete tumour resection is not considered to be feasible without substantial risk or morbidity, or if a patient with a surgical option refuses surgery.

   * Since there is no standard effective chemotherapy for patients with NF1 and PN, subjects may be treated on this trial without having received prior medical therapy directed at their PN. For Phase 2 Cohort B in subjects with NF-1 related OPGs at least two prior standard therapies need to have been received.
   * Subjects who have received previous investigational agents or biologic therapy except a prior MEK inhibitor are eligible for enrollment. At least 4 weeks must have elapsed since receiving medical therapy directed at the PN. Patients who received prior medical therapy for their PN must have recovered from the acute toxic effects of all prior therapy to ≤ grade 1 CTCAEv4 before entering this study.
   * Growth factors that support platelet or white cell number or function must not have been administered within the past 7 days.
   * At least 6 weeks must have elapsed prior to enrollment since the patient received any prior radiation therapy.
5. Performance status: Patients ≥ 16 years of age must have a Karnofsky performance level of ≥70%, and children < 16 years old must have a Lansky performance of ≥70% (Error! Reference source not found.). Patients who are wheelchair bound because of paralysis secondary to a plexiform neurofibroma should be considered ambulatory when they are up in their wheelchair. Similarly, patients with limited mobility secondary to need for mechanical support (such as an airway PN requiring tracheostomy or CPAP) will also be considered ambulatory for the purpose of the study.
6. Haematological Function: Patients must have an absolute neutrophil count ≥1500/µl, haemoglobin ≥9g/dl, and platelet ≥100,000/µl.
7. Hepatic Function: Patients must have bilirubin within 1.5 x the upper limit of normal for age, with the exception of those with Gilbert syndrome, and AST/ALT within ≤ 2.5 x upper limit of normal.
8. Renal Function: Patients must have a creatinine clearance or radioisotope GFR ≥60ml/min/1.73 m2 or a normal serum creatinine based on age described in the table below.

   Age (years) Maximum Serum Creatinine (mg/dL) age ≤5: 0.8 5<age≤10: 1.0 10<age≤15: 1.2 age>15: 1.5
9. Cardiac Function: Normal ejection fraction (ECHO) ≥ 55%, or institutional normal value (if a range is given then the upper value of the range will be used); QTcF ≤450 msec.
10. Adequate Blood Pressure defined as:

    A blood pressure (BP) ≤ the 95th percentile for age, height, and gender. Adequate blood pressure can be achieved using medications for treatment of hypertension.
11. Informed Consent: Diagnostic or laboratory studies performed exclusively to determine eligibility for this trial must only be done after obtaining written informed consent from all patients or their legal guardians (if the patient is <16 years old). When appropriate, paediatric patients will be included in all discussions and appropriate assent taken.
12. Willingness to avoid excessive sun exposure and use adequate sunscreen protection if sun exposure is anticipated.
13. Willingness to avoid the ingestion of grapefruit and Seville oranges (as well as other products containing these fruits, e.g. grapefruit juice or marmalade) during the study.

Exclusion Criteria:

1. Pregnant or breast-feeding females are excluded due to potential risks of foetal and teratogenic adverse events of an investigational agent. Pregnancy tests must be obtained prior to enrolment on this study for girls of reproductive potential. The need to commence pregnancy testing will be at the discretion of the treating physician to facilitate taking in to account factors such as precocious puberty, endocrine status and medications which can affect pubertal status. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. Abstinence is an acceptable method of birth control.
2. Known severe hypersensitivity to selumetinib or any excipient of selumetinib or history of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib.
3. Recent major surgery within a minimum of 4 weeks prior to starting study treatment, with the exception of surgical placement for vascular access.
4. Phase I: Patients who anticipate the need for surgical intervention within the first three cycles (3 months), as surgical intervention during the period of DLT evaluation may affect analysis of adherence and/or make the subject in-evaluable.

   Phase II: Patients who anticipate the need for surgical intervention of the target PN within the first eight cycles (8 months), as surgical intervention during the period may affect analysis of response and may make the subject in-evaluable.
5. An investigational agent within the past 28 days.
6. Any unresolved chronic toxicity with toxicity ≥ CTCAE Grade 2 from previous anti-cancer therapy, except for alopecia.
7. Ongoing radiation therapy, chemotherapy, hormonal therapy directed at the tumour, immunotherapy, or biological therapy.
8. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
9. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
10. Inability to swallow capsules, since capsules cannot be crushed or broken.
11. Inability to undergo MRI and/or contraindication for MRI examinations following the MRI protocol. Prosthesis or orthopaedic or dental braces that would interfere with volumetric analysis of target PN on MRI.
12. Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
13. Prior treatment with selumetinib or another specific MEK1/2 inhibitor.
14. Evidence of an optic glioma (progressive OPG allowed in Phase 2), malignant glioma, malignant peripheral nerve sheath tumour, or other cancer requiring treatment with chemotherapy or radiation therapy.
15. Patients should not take any supplementation with Vitamin E.
16. Patients not achieving adequate blood pressure in spite of antihypertensive therapy for control of blood pressure.
17. Cardiac Function:

    1. Known inherited coronary disease
    2. Symptomatic heart failure (NYHA Class II-IV prior or current cardiomyopathy, or severe valvular heart disease)
    3. Prior or current cardiomyopathy
    4. Severe valvular heart disease
    5. History of atrial fibrillation
18. Ophthalmologic conditions:

    1. Current or past history of central serous retinopathy
    2. Current or past history of retinal vein occlusion

    <!-- -->

    1. Patients with controlled known glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) and are not experiencing pain related to the glaucoma, may be eligible after discussion with the PI.
    2. Subjects with any other significant abnormality on ophthalmic examination (performed by an ophthalmologist) should be discussed with the PI for potential eligibility
    3. Ophthalmological findings secondary to optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) or long-standing orbito-temporal PN (such as visual loss, strabismus) will NOT be considered a significant abnormality for the purposes of the study
19. Clinical judgement by the investigator that the patient should not participate in the study.
20. While not an exclusion criterion, unless considered clinically indicated, patients should avoid taking other additional non-study medications that may interfere with the study medication. In particular, patients should avoid medications that are known to either induce or inhibit the activity of hepatic microsomal isoenzymes CYP1A2, CYP2C19 and CYP3A4, as this may interfere with the metabolism of selumetinib.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Phase 1: To evaluate the Maximum Tolerated Dose | 6 months
  Phase 1: Definition of the maximum tolerated dose using number of participants with treatment related adverse events as assessed by CTCAEv4.0
Phase 2: Objective response rate in NF1 inoperable plexiform neurofibroma and optic pathway glioma | 2 years
  Phase 2:To evaluate the objective response rate of children (≥3 and ≤ 18 years old) with NF1 and inoperable plexiform neurofibroma using 3D volumetric analysis.
Best Objective response rate in NF1 related optic pathway gliomas | 2 years
  To evaluate the best objective response rate (including MR, PR and CR) of children (≥3 and ≤ 18 years old) with NF1 related optic pathway glioma using 2D assessment of tumour size.

SECONDARY OUTCOMES:
Cardiac Function - fractional shortening | 5 years
  Number of patients with changes in changes from baseline in ejection fraction as assessed by echocardiogram.
Cardiac Function - QTc | 5 years
  Number of patients with changes from baseline in QTc as assessed by electrocardiogram.
Retinal detachment. | 5 years
  Number of participants with evidence of treatment related retinal detachment as per CTCAE v4.
Treatment related Adverse Events | 5 years
  Number of participants with Treatment- Related Adverse events as assessed by CTCAEv4.0.
Pharmacokinetics of selumetinib. Phase 1 only | 6 months
  Calulation of Area Under the Curve (AUC) tests to test exposure to the drug over time. AUC will be calculated at Day 1 and at steady state (Day 27/28)
Pharmacokinetics of selumetinib. Phase 1 only | 6 months
  Calculation of Time to reach peak concentration (Tmax) at day 1 and at steady state (Day 27/28)
Pharmacokinetics of selumetinib. Phase 1 only | 6 months
  Calculation of Peak concentration (Cmax) at day 1 and at steady state (Day 27/28)
Pharmacokinetics of selumetinib. Phase 1 only | 6 months
  Calculation of clearance of the drug from the blood after oral administration (CL/F) on day 1 and at steady state (D27/28)
Time to progression - plexiform neurofibromas | 5 years
  Definition of time to progression of plexiform neurofibromas as assessed by volumetric measurement.
Time to progression - optic pathway gliomas | 5 years
  Definition of time to progression as defined by changes from baseline using 2 dimensional assessment of tumour size
Pain Evaluation - self reported changes | 3 years
  Number of participants with a change from baseline as assessed by Numerical Scale Rating
Pain Evaluation- Medication | 3 years
  Number of participants with a change from baseline in pain medication as assessed by the pain medication survey.
Evaluation of effect on disfigurement | 3 years
  Photography evaluation (imaging including standardised imaging and 3D photography where available) to provide measurement (metric system eg cm) of change from baseline in size of deformity caused by plexiform neurofibroma.
Quality of Life Evaluation | 3 years
  Number of participants with a change from baseline in quality of life using the PedsQL assessment.
Evaluation of Visual Function in NF1 related optic pathway glioma | 3 years
  To determine the effect of selumetinib on visual function in subjects with NF1 related optic pathway glioma using the visual function assessments outlined by the Response Evaluation in Neurofibromatosis and Schwanomatosis (REiNS) criteria
Physical functioning endurance | 3 years
  Number of participants with a change in physical function as assessed using the 6 minute walk-run test.
Evaluation of clinically stable NF1 related optic pathway glioma | 5 years.
  To determine the effect of selumetinib on stable NF1 related optic pathway gliomas and other gliomas for subjects whose primary indication for treatment is a progressive plexiform neurofibroma using evaluation of CNS MRI imaging
Functional Outcome of patients with Plexiform Neurofibromas affecting the airway - PFT | 3 years
  Number of participants who have a change from baseline in their pulmonary function as assessed by pulmonary function testing.
Functional outcome of participants with plexiform neurofibromas affecting the airway - sleep studies | 3 years
  Number of participants who have a change from baseline, in their airway function as assessed by sleep studies.
Functional Outcome of patients with Plexiform Neurofibromas affecting motor strength - grooved pegboard test | 3 years
  Number of participants who have a change from baseline in their muscle strength using grooved pegboard test.
Functional Outcome of patients with Plexiform Neurofibromas affecting motor strength.- MRC grading of strength | 3 years
  Number of participants who have a change from baseline in their muscle strength using medical research council (MRC) grading system.
Functional Outcome of patients with Plexiform Neurofibromas affecting motor strength. | 3 years
  Number of participants who have a change from baseline in their muscle strength using leg length evaluation.
Functional Outcome of patients with plexiform neurofibromas which affect mobility. | 3 years
  number of participants who have a change from baseline in the patient reported outcome score (numerical scale rating) of mobility. PROMIS forms will be used.
Functional Outcome of patients with plexiform neurofibromas which affect bladder and bowel function. | 3 years
  Measurement of bladder and bowel function using patient reported outcomes (tick box questionnaire) covering urgency, frequency, dysuria, constipation and incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Darren Hargrave, MB Bch, Principal Investigator — Great Ormond Street Hospital NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Great Ormond Street Hospital NHS Foundatin Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dombi E, Baldwin A, Marcus LJ, Fisher MJ, Weiss B, Kim A, Whitcomb P, Martin S, Aschbacher-Smith LE, Rizvi TA, Wu J, Ershler R, Wolters P, Therrien J, Glod J, Belasco JB, Schorry E, Brofferio A, Starosta AJ, Gillespie A, Doyle AL, Ratner N, Widemann BC. Activity of Selumetinib in Neurofibromatosis Type 1-Related Plexiform Neurofibromas. N Engl J Med. 2016 Dec 29;375(26):2550-2560. doi: 10.1056/NEJMoa1605943. PMID 28029918
- [Background] Banerjee A, Jakacki RI, Onar-Thomas A, Wu S, Nicolaides T, Young Poussaint T, Fangusaro J, Phillips J, Perry A, Turner D, Prados M, Packer RJ, Qaddoumi I, Gururangan S, Pollack IF, Goldman S, Doyle LA, Stewart CF, Boyett JM, Kun LE, Fouladi M. A phase I trial of the MEK inhibitor selumetinib (AZD6244) in pediatric patients with recurrent or refractory low-grade glioma: a Pediatric Brain Tumor Consortium (PBTC) study. Neuro Oncol. 2017 Aug 1;19(8):1135-1144. doi: 10.1093/neuonc/now282. PMID 28339824